CLINICAL TRIAL: NCT00522977
Title: Echo-Cardiographic Assessment of Cardiovascular Characteristics During Pregnancy and Postpartum Periods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Other Study IDs: BLOND1CTIL
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Pregnancy
Keywords: Myocardial strain; Myocardial function; Pregnancy; Postpartum; Echocardiography; Myocardial adaptation to pregnancy; Systolic function; Diastolic function

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this echocardiographic study is to restudy the longitudinal changes in cardiac size and function during and after pregnancy in healthy women using relatively new parameters of systolic and diastolic function as well as classical measures of left ventricle (LV) function using contemporary echocardiographic machines.

We, the researchers at Hillel Yaffe Medical Center, will assess diastolic function and its possible relation to shortness of breath.

DETAILED DESCRIPTION:
A comprehensive echocardiographic study of the heart will be conducted in the first, second and third trimesters of pregnancy and 3 months postpartum.

Determination of left ventricular dimensions, transvalvular Doppler flow, ejection fraction, stroke volume, cardiac output, pulmonary vein flow, tissue Doppler, flow propagation, global and segmental strain parameters, timing of peak strain and various parameters of diastolic function will be obtained.

From these data normal values for various stages of pregnancy will be determined as well as range for changes expected during longitudinal follow-up will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* First trimester of a normal pregnancy
* Normal baseline echocardiogram

Exclusion Criteria:

* Pregnancy with more than one fetus.
* Any hemodynamically significant cardiac condition
* Any known systemic disease
* Poor quality echocardiogram

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy women in first trimester of pregnancy.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-08; Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David S Blondheim, MD, Principal Investigator — Hillel Yaffe Medical Center; Asnat Walfisch, MD, Principal Investigator — Hillel Yaffe Medical Center; Mordechai Hallak, Prof., Study Chair — Hillel Yaffe Medical Center; Avraham Shotan, MD, Study Director — Hillel Yaffe Medical Center; Kazatzker Mark, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel